CLINICAL TRIAL: NCT03635060
Title: Distraction Osteogenesis for Distal Radius Fractures vs. Volar Plating
Acronym: DORSAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Patrick Henry, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DORSAL
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorsal Bridge Plating (Active Comparator): The intervention is surgery with dorsal distraction plating with or without any additional fragment specific fixation.
  Interventions: Procedure: Dorsal Bridge Plating
- Volar Locking Plating (Active Comparator): The intervention is surgery with open reduction and internal fixation with non-spanning fixation.
  Interventions: Procedure: Volar locking plating

INTERVENTIONS:
Procedure: Dorsal Bridge Plating — This study will be a pilot randomized control trial that will focus on treating patients with the described fracture pattern either with dorsal distraction plating with or without any additional fragment specific fixation or standard open reduction internal fixation.
  Arms: Dorsal Bridge Plating
Procedure: Volar locking plating — This study will be a pilot randomized control trial that will focus on treating patients with the described fracture pattern either with dorsal distraction plating with or without any additional fragment specific fixation or standard open reduction internal fixation.
  Arms: Volar Locking Plating

SUMMARY:
Optimal fixation for highly comminuted distal radius fractures with metadiaphyseal extension remains to be a major treatment challenge for orthopaedic surgeons. The purpose of this study is to determine the safety, feasibility and sample size estimations for a larger, definitive study comparing functional outcomes of patients treated with dorsal distraction plate fixation with or without fragment specific fixation to standard open reduction internal fixation in highly comminuted distal radius fractures (subtypes AO.23-C2 and AO.23-C3). The study design will be a pilot randomized control trial. Fracture pattern eligibility will be determined by consensus agreement between two fellowship trained upper extremity specialists. The primary outcome measure will be the QuickDASH score. Secondary outcome measures include wrist range of motion, grip strength, Visual Analog Scale pain scale, Short Form SF-12, and EQ-5D. Ultimately, this study will lead to a larger randomized control trial and result in improvement in the care and treatment of patients with these challenging injuries.

DETAILED DESCRIPTION:
Distal radius fractures are the most common long bone fractures and the incidence appears to be increasing worldwide. They have been found to account for approximately 17% of all fracture related emergency department visits. These types of injuries have a bimodal age distribution. The first cohort consists of elderly patients with lower to moderate energy injuries secondary to osteoporosis, and the second cohort consists of young patients involved in high energy traumas.

Surgical treatment for distal radius fractures varies, as there are numerous techniques for fixation. The goals of fixation are anatomic reduction and stability, as this has been shown to result in improved chances for functional recovery. The use of volar distal radius locking plates has become the standard for treatment of the majority of low-energy distal radius fractures. However, adequate fixation for high energy comminuted fractures with or without metadiaphyseal extension remains a major treatment challenge. Severely comminuted articular fractures are problematic in terms of obtaining an adequate reduction and/or stabilization by the standard periarticular plate. It is in this light that the dorsal distraction plate can serve as an improved fixation device by allowing comminuted articular fragments reduce under ligamentotaxis. In addition, periarticular plate fixation cannot address proximal comminution. Furthermore, the use of external fixation has fallen out of favour due to the high complication rate associated with pin track infections resulting in loosening and loss of reduction. It has been reported that highly comminuted distal radius fractures are associated with a 52% to 63% complication rate when treated with external fixation. Recently, there has been increased use of dorsal distraction plating for these types of injuries however, the literature to date is quite limited. Unlike external fixation, the bridge plate can be left in place for an extended period of time without the risk of the aforementioned complications.

Burke and Singer were the first to describe use of internal distraction plating for treatment of comminuted, displaced distal radius fractures in 1998. Since then, the literature on outcomes after dorsal distraction plating has been limited to retrospective reviews except for one prospective series by Ruch et al in 2005. The rationale for an internal spanning plate is multifactorial. Firstly, it is an extremely stable construct and more rigid than an external fixator. Secondly, due to the extensive time required for bone healing (approximately 12 weeks), in these injuries, the internal distraction plate can remain in situ until full union has completed. Lastly, this method allows for early weight bearing and transfer in polytraumas patients with pelvic or lower extremity injuries.

Despite the increasing use of dorsal distraction plating for these types of injuries, there has not been a proper analysis comparing dorsal distraction plating to standard open reduction internal fixation volar plating. Furthermore, most of the studies in the literature have varied in terms of outcome assessment. Much of the current literature has found that this type of fixation results in restoration of functional range of motion with minimal complications rates. More detailed information regarding outcomes following this type of fixation may help improve functional outcomes post-injury as well as improve mobilization in polytrauma patients. Using a comprehensive approach to evaluating patients, the investigators aim to initially perform a retrospective case series study of patients treated with dorsal distraction plating versus open reduction internal fixation volar plating. Once completed, the investigators plan to perform a pilot randomized control trial comparing the same groups described previously for AO.23-C2 and AO.23-C3 distal radius fractures.

The aim of this study is to evaluate the use of dorsal distraction plating alone or combined with any other fragment specific fixation in the treatment of severely comminuted distal radius fractures with metadiaphyseal extension (AO.23-C2 and AO.23-C3) and compare outcomes to those treated with open reduction internal fixation.

The investigators hypothesize that highly comminuted distal radius fractures with metadiaphyseal extension treated with dorsal distraction plating result in restoration of function as well as improved outcomes compared to those treated with standard open reduction internal fixation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 years
* Diagnosed with unilateral or bilateral, open or closed, severely comminuted distal radius fractures (fracture classification of AO.23-C2 and AO.23-C3)
* Scheduled to undergo surgery

Exclusion Criteria:

* Previous wrist injuries or surgery that would compromise performance of either procedure.
* Surgery delayed beyond 21 days from injury.
* Significant medical comorbidities.
* Neurologic injury causing paralysis of affected arm.
* Those unable to attend follow up and comply with the post-operative protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
QuickDASH | primary outcome assessed at 1 year following surgery (survey done at each followup starting at week 6)
  It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level.

SECONDARY OUTCOMES:
Change in Patient-Related Wrist Evaluation | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following surgery
  The Patient Related Wrist Evaluation is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. Developed in 1998 for clinical assessment and is used for specific wrist problems. It is one of the reliable upper extremity outcome instruments.
EQ-5D | 6 weeks, 3 months, 6 months, and 1 year following surgery
  A standardized instrument for measuring generic health status. The health status measured with EQ-5D is used for estimating preference weight for that health status, then by combining the weight with time, quality-adjusted life year (QALY) can be computed. QALYs gained is used as an outcome in cost-utility analysis which is a type of economic evaluation that compares the benefit and cost of health care programs or interventions.

OTHER OUTCOMES:
Range of Motion | 3 months, 6 months, and 1 year following surgery
  Range of motion will be recorded including flexion/extension/supination/pronation.
Grip Strength | 6 weeks, 3 months, 6 months, and 1 year following surgery
  Grip strength for injured and non-injured limbs measured using standard dynamometer.
Anterior-posterior x-rays | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following surgery
  Anterior-posterior x-rays to assess radial inclination, volar tilt, degree of radiocarpal arthritis, radial length, tear drop angle, and articular step-off.
Lateral x-rays | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following surgery
  Lateral x-rays to assess radial inclination, volar tilt, degree of radiocarpal arthritis, radial length, tear drop angle, and articular step-off.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No